CLINICAL TRIAL: NCT00839098
Title: Powered Seating Function Usage Among Veterans - Compliance and Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B6591-R
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Use of Power Wheelchairs and Power Seat Functions
Keywords: power wheelchairs; assistive technology; rehabilitation
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (No Intervention): Control Group
- Instruction Group (Experimental): Instruction Group
  Interventions: Other: Instruction Group: Power seat function usage instruction- verbal and written instruction
- Instruction and Virtual Coach Group (Experimental): Instruction and Virtual Coach Group
  Interventions: Other: Instruction and Virtual Coach Group: Power seat function usage instruction- verbal, written, and virtual coach

INTERVENTIONS:
Other: Instruction Group: Power seat function usage instruction- verbal and written instruction — Subjects assigned to the Intervention Group will be assigned to an Intervention Group Clinician. The Intervention Group Clinicians will provide the same training as the Control Group Clinicians, with the addition of discussing the Veteran's activity and seating function usage data, reviewing and providing a study pamphlet and compact disk as a reference guide on use of power seat functions.
  Arms: Instruction Group
Other: Instruction and Virtual Coach Group: Power seat function usage instruction- verbal, written, and virtual coach — Subjects assigned to the Instruction & Virtual Coach Group will be assigned to an Intervention Group Clinician and will receive the same training and instructional materials as the Instruction Group. Subjects will also be instructed in use of the virtual coach system, which will be active during the in-home usage periods to provide personalized feedback. As the Virtual Coach is a dynamic intelligent system, it will adjust its coaching to the needs of the individual. For example, if the person is compliant, the Virtual Coach will give positive feedback and then gradually transition to operating quietly in the background. If a person is not fully compliant, it will alter feedback modes (e.g., verbal cues, auditory tones, visual cues) and timing to attempt to increase compliance.
  Arms: Instruction and Virtual Coach Group

SUMMARY:
The purpose of this randomized control study is to evaluate the use of electric powered wheelchairs and powered seating function patterns of Veterans to determine how usage patterns relate to activity, participation, and seating discomfort. In addition, it will be determined if a training program or a training program with a virtual coach will improve compliance of clinical practice guidelines for pressure relief, upper limb preservation, and discomfort management. The virtual coach is a portable, programmable intelligent reminder designed to enhance a person's use of their power wheelchair and power seat functions.

DETAILED DESCRIPTION:
This is a randomized control trial evaluating power seat function usage among 3 groups: 1) standard of care- verbal instruction 2) verbal and written instruction and 3) same as #2 with addition of virtual coach. This study will be conducted in two phases. Phase I data will be collected for 8 weeks, during the time period that the subject is awaiting for delivery of their personal electric powered wheelchair (EPW) with powered seat functions. Phase II data will be collected for a total of 4 weeks, after the subject receives their personal wheelchair. During Phase I, Visit I, subjects will be fitted for a study EPW with powered seat functions. All subjects will be provided with the "standard of care" training on driving of the wheelchair and usage of the power seating functions. Subjects will be instructed to go about their daily activities as they normally would, while the instrumented wheelchair will track their usage of the wheelchair and seating habits. Phase I, Visit II-IV, subjects will be randomized into one of three study groups: Control Group; Instruction Group; and Instruction & Virtual Coach Group. Subjects assigned to the Control Group will receive 'standard of care.' Subjects assigned to the Intervention Group will receive the "standard of care" and additional written instructional materials and feedback regarding activity and wheelchair usage. Subjects assigned to the Instruction & Virtual Coach Group will receive the same training and instructional materials as the Intervention Group. This group will also be instructed in use of the virtual coach system, which will be active during the in-home usage periods to provide personalized feedback. Phase II will involve mounting a wheelchair and seat function usage datalogger to the subject's personal wheelchair over a period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older.
* A power wheelchair with power seat functions must be recommended as medically necessary by a qualified clinician with ATP credential or board certified in physical medicine and rehabilitation from the VAPHS Wheelchair and Seating Clinic or the Center for Assistive Technology.
* Subjects must be able to be properly fitted with one of the study EPWs; 18" or 20" seat widths will be available. Cushions and backrests will be made available to meet subject's clinical needs.
* Subject's home must be accessible to accommodate use of a power w/c.
* Subject must be determined to be fully capable of examining his/her sitting surface daily for redness or pressure ulcers or if not that another individual can be designated as able and willing to-do this.

Exclusion Criteria:

* Subjects who have active pelvic, gluteal or thigh wounds or who have had a pressure ulcer in these regions within the past 30 days. (They may be worsened by prolonged sitting).
* Subjects who report more than 5 days of hospitalization in the previous month. (They may not spend enough time using an EPW with powered seating functions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rory A. Cooper, PhD, Principal Investigator — Director, Center of Excellence for Wheelchairs and Related Technology
Locations (1):
- VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Instruction Group | Instruction and Virtual Coach Group
Started | 3 | 12 | 13
Completed | 1 | 11 | 6
Not Completed | 2 | 1 | 7
Not completed — Withdrawal by Subject | 2 | 1 | 7

BASELINE CHARACTERISTICS:
Population: The average age of the participants was 53.2 years old (+/- 14.0 years old). Twelve out of 28 were female (42.9%). Two of the participants were veterans, and one of them was recruited from VA Wheelchair Seating clinic.
  Arm 1 (control group) was removed from the study through IRB modification because of difficulties in recruiting participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Instruction Group | Instruction and Virtual Coach Group | Total
Number analyzed (Participants) | 3 | 12 | 13 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 11 | 9 | 23
  >=65 years | 0 | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: Years of age] | 47.0 (19.9) | 53.4 (9.1) | 54.5 (17.0) | 53.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 5 | 12
  Male | 1 | 7 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 3 | 12 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Compliance Rate
Description: Compliance rate is a measure of compliance with the recommendation of using powered seating functions (moderate or maximum range of tilt, at least once every hour, for 2 minutes). The participant had to follow the recommended position, duration, and frequency to be considered as compliant and performed successful repositioning exercise. The compliance rate of a participant was the number of successful repositioning exercise divided by the sum of the number of successful repositioning exercise and missed repositioning exercise. The result of the difference between the baseline and week 7-8 (last 2 weeks) was shown here.
Time Frame: Every 2 weeks for 8 weeks following acquisition of wheelchair
Population: Only the data of the participants who completed the study protocol and use the wheelchair were included in the data analysis.
Measure: Mean (Standard Deviation); unit: Percentage of participants' compliance
Groups:
- Arm 1: Control Group: Arm 1 (control group) was removed from the study through IRB modification because of difficulties in recruiting participants.
- Arm 2: Instruction Group: Participants received: meeting with a clinician once every two weeks, and educational materials (reminder cards, pamphlet, and video CD).
- Arm 3: Instruction + VSC Group: Participants received: meeting with a clinician once every two weeks, and educational materials (reminder cards, pamphlet, and video CD), and timely alert to remind and guide powered seating function usage delivered by the VSC installed on the study wheelchair.
Arm/Group | Arm 1: Control Group | Arm 2: Instruction Group | Arm 3: Instruction + VSC Group
Number analyzed (Participants) | 0 | 10 | 6
Percentage of participants' compliance |  | 8.9 (15.9) | 39.7 (23.5)
Statistical Analysis 1: Comparison: Arm 2: Instruction Group vs Arm 3: Instruction + VSC Group; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Questionnaire Responses: Tool for Assessing Wheelchair Discomfort (TAWC)
Description: General Discomfort Assessment (GD) and Discomfort Intensity Rating (DI) are two sub-scales of TAWC. Higher scores indicate greater discomfort. GD consists of 8 discomfort statements and 5 comfort statements. The statements are rated on a seven point Likert scale, from strongly disagree to strongly agree of points from 1-7 (total score: 13-91). DI includes seven body areas (back, neck, buttocks, legs, arms, feet, and hands) and overall discomfort level, rated for a degree of discomfort intensity on a scale of 0 (no discomfort) to 10 (severe discomfort). Space is also included for the user to list additional body areas. DI scores may range from 0 to more than 80, depending on whether the participant reported additional areas of discomfort. Although GD and DI were measured daily, the data were average for each two-week period. The average GD and DI of the difference between the baseline and week 7-8 (last 2 weeks) were shown here.
Time Frame: Every 2 weeks for 8 weeks following acquisition of wheelchair
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Control Group | Arm 2: Instruction Group | Arm 3: Instruction + VSC Group
Number analyzed (Participants) | 0 | 10 | 6
units on a scale
  General Discomfort: Difference |  | 4.6 (7.5) | -7.4 (16.9)
  Discomfort Index: Difference |  | 1.8 (10.0) | -12.1 (13.6)
Statistical Analysis 1: Comparison: Arm 2: Instruction Group vs Arm 3: Instruction + VSC Group; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Questionnaire Responses: Psychological Impacts of Assistive Devices Scale
Description: This tool is to measure perceived psychological impact of using an assistive device. It consists of three subscales, Competence (12 items), Adaptability (6 items), and Self-esteem (8 items). Each item is scored on a likert scale from -3 (decreases) to + 3 (increases). The total score is the sum of all 26 items, ranging from -78 to 78. A higher positive score indicates more positive impact. A negative score indicates negative impact. The differences between the measurements taken at the end of 2nd week (end of baseline) and the end of 8th week (end of intervention period) are reported here to show the intervention effect.
Time Frame: At the end of every two weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Control Group | Arm 2: Instruction Group | Arm 3: Instruction + VSC Group
Number analyzed (Participants) | 0 | 10 | 6
units on a scale |  | 11.1 (17.7) | -8.4 (15.6)
Statistical Analysis 1: Comparison: Arm 2: Instruction Group vs Arm 3: Instruction + VSC Group; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Questionnaire Responses: Independence in Community
Description: This outcome was measured in three aspects: Physical Independence, Cognitive Independence, and Mobility, using the three of the subscales of Craig Handicap Assessment and Reporting Technique Scale. The scores of each subscale has to be calculated with specific formula and weight based on the manual. The range of each subscale score are: Physical Independence: 28-100; Cognitive Independence: 15-100; and Mobility: 16-100. A higher score indicates greater independence. The analyzed results of the difference between the measurements at the end of 2nd week and 8th week were shown here.
Time Frame: At the end of 2nd (end of baseline) week and 8th week (end of intervention period) following acquisition of wheelchair
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Control Group | Arm 2: Instruction Group | Arm 3: Instruction + VSC Group
Number analyzed (Participants) | 0 | 10 | 6
units on a scale
  Phy. Independence: Difference |  | 9.5 (55.6) | 8.6 (49.2)
  Cog. Independence: Difference |  | 19.3 (38.2) | -11.7 (18.3)
  Mobility: Difference |  | 0 (22.5) | 0.5 (17.2)
Statistical Analysis 1: Comparison: Arm 2: Instruction Group vs Arm 3: Instruction + VSC Group; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Frequency of Power Seat Function Usage
Description: Frequency of power seat function usage was measured by the number of times of changing tilt and recline angles averaged by the duration that the participant occupied the wheelchair per day. The results of the difference between the baseline and week 7-8 (last 2 weeks) were shown here.
Time Frame: Every 2 weeks for 8 weeks following acquisition of wheelchair
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: times/hour
Arm/Group | Arm 1: Control Group | Arm 2: Instruction Group | Arm 3: Instruction + VSC Group
Number analyzed (Participants) | 0 | 10 | 6
times/hour
  Freq of mod & max tilt (times/hr): Difference |  | .51 (2.52) | 0.03 (2.51)
  Freq of mod & max recline (times/hr): Difference |  | -0.43 (1.36) | 0.09 (0.15)
Statistical Analysis 1: Comparison: Arm 2: Instruction Group vs Arm 3: Instruction + VSC Group; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Power Wheelchair Usage
Description: Power wheelchair usage was measured by the sum of distances that the power wheelchair traveled (km) divided by the duration of the wheelchair being occupied a day (hr). The result of the difference between the baseline and week 7-8 (last 2 weeks) was shown here.
Time Frame: Every 2 weeks for 8 weeks following acquisition of wheelchair
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: km/hour
Arm/Group | Arm 1: Control Group | Arm 2: Instruction Group | Arm 3: Instruction + VSC Group
Number analyzed (Participants) | 0 | 10 | 6
km/hour |  | 0.17 (0.45) | -0.04 (0.08)
Statistical Analysis 1: Comparison: Arm 2: Instruction Group vs Arm 3: Instruction + VSC Group; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — P values below 0.05 were considered statistically significant in this study

7. Primary Outcome: Wheelchair Occupancy
Description: Wheelchair occupancy was measured by the sum of duration that the seat of the wheelchair was occupied. The results of the difference between the baseline and week 7-8 (last 2 weeks) were shown here.
Time Frame: Every 2 weeks for 8 weeks following acquisition of wheelchair
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm 1: Control Group | Arm 2: Instruction Group | Arm 3: Instruction + VSC Group
Number analyzed (Participants) | 0 | 10 | 6
hours |  | -.07 (1.9) | -0.4 (1.8)
Statistical Analysis 1: Comparison: Arm 2: Instruction Group vs Arm 3: Instruction + VSC Group; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Control Group | Instruction Group | Instruction and Virtual Coach Group
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/3 | 0/12 | 0/13

LIMITATIONS AND CAVEATS:
It was difficult to recruit power wheelchair users to participate in the study. Participants withdrew from the study because the study wheelchair could not meet their needs, or they could not use the Virtual Seating Coach independently.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No